CLINICAL TRIAL: NCT00522548
Title: Gastrointestinal Adverse Effect Outcomes of De Novo African American Kidney Transplant Recipients Treated With Tacrolimus, Corticosteroids and Mycophenolate Mofetil or Enteric Coated Mycophenolate Sodium
Brief Title: Myfortic or CellCept Gastrointestinal Effects in African American Kidney Recipients
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: enrollment halted in order to have all patients complete follow-up by Jan 2011
Sponsor: University of Pennsylvania (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Roy D. Bloom, MD, Medical Director, Penn Kidney/Pancreas Transplant Program, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CERL080A-US49
Record Dates: First submitted 2007-08-27; First posted 2007-08-29 (Estimated); Results first posted 2018-01-23 (Actual); Last update posted 2018-01-23 (Actual); Status verified 2017-12

CONDITIONS: Transplants and Implants
Keywords: African American; Kidney Transplant
MeSH Terms: interventions — Mycophenolic Acid

STUDY DESIGN:
Intervention Model Description: This study consisted of 2 parallel active comparator arms.
Masking Description: Masking description is not applicable since no masking was used in this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Enteric coated mycophenolate sodium (Active Comparator): Patients in this group will receive Myfortic (enteric-coated mycophenolate sodium) at a target dose of 720 mg orally twice daily for 6 months after transplant.
  Interventions: Drug: Enteric coated mycophenolate sodium
- Mycophenolate mofetil (Active Comparator): Patients in this group will receive CellCept (mycophenolate mofetil) or its generic equivalent manufactured by Sandoz, at a target dose of 1000 mg orally twice daily for 6 months after transplant.
  Interventions: Drug: Mycophenolate mofetil

INTERVENTIONS:
Drug: Enteric coated mycophenolate sodium — Patients in this group will receive Myfortic (enteric-coated mycophenolate sodium) in combination with Thymoglobulin (rabbit Anti-thymocyte globulin) induction immunosuppression, Prograf (tacrolimus) or its generic equivalent, and corticosteroid immunosuppression.
  Other Names: Myfortic
  Arms: Enteric coated mycophenolate sodium
Drug: Mycophenolate mofetil — Patients in this group will receive CellCept (mycophenolate mofetil) or its generic equivalent formulation manufactured by Sandoz, in combination with Thymoglobulin (rabbit Anti-thymocyte globulin) induction immunosuppression, Prograf (tacrolimus) or its generic equivalent, and corticosteroid immunosuppression.
  Other Names: CellCept
  Arms: Mycophenolate mofetil

SUMMARY:
Myfortic (enteric-coated mycophenolate sodium) has been shown to have similar effectiveness to CellCept (mycophenolate mofetil) in preventing rejection in kidney transplant recipients. However, enteric coated mycophenolate sodium has been thought to possibly be associated with fewer gastrointestinal side effects. Mycophenolate mofetil and enteric coated mycophenolate sodium pharmacokinetics (how the drug is absorbed and broken down) have not been well-studied in African American kidney transplant recipients. The investigators are interested in studying enteric coated mycophenolate sodium and mycophenolate mofetil pharmacokinetics and gastrointestinal side effects in African American kidney transplant recipients.

DETAILED DESCRIPTION:
African American patients often experience more gastrointestinal (GI) complications after kidney transplant than Caucasian patients. In addition, African American kidney transplant recipients also experience a higher incidence of acute rejection and have worse outcomes compared with all other ethnic groups. Reasons accounting for these differences are not well understood.

In light of the increased risk of GI complications in African American patients, we will compare in a pilot study, different regimens (described below) that we commonly use in our clinical practice in this population. As part of this study, patients will also fill out a GSRS survey at specified time points to help describe gastrointestinal side effects after transplant.

Pharmacokinetic studies (studies looking at how the drugs are absorbed and broken down) for mycophenolate mofetil or enteric coated mycophenolate sodium have largely been performed in Caucasian populations. There is little information available in African-American patients. This is particularly concerning in the face of the worst clinical outcomes observed after transplantation in African American kidney transplant recipients.

Comparisons: Patients will be randomized to one of two groups

* Group 1: Myfortic (enteric-coated mycophenolate sodium) in combination with Prograf (tacrolimus) or its generic equivalent and corticosteroids
* Group 2: CellCept (mycophenolate mofetil) or its generic equivalent manufactured by Sandoz in combination with Prograf (tacrolimus) or its generic equivalent and corticosteroids

Since toxicity of mycophenolate mofetil and enteric coated mycophenolate sodium may be influenced by pharmacokinetics (studies that look at how the drugs are absorbed and broken down) of these respective drugs, we will compare the pharmacokinetics of enteric coated mycophenolate sodium and mycophenolate mofetil in a subset of patients. This pharmacokinetic data may have the additional valuable benefit of helping to optimize dosing parameters for mycophenolate mofetil and enteric coated mycophenolate sodium in African American kidney transplant patients in the future.

ELIGIBILITY:
Inclusion Criteria:

* Recipients of a deceased donor or living donor kidney transplant
* Recipients of age greater than 18 years but less than 76 years
* African Americans (self-reported patients of Black African descent who live in the United States)
* Willingness to participate in a randomized, clinical trial, as indicated by signed informed consent
* Patients with a history of gastrointestinal complications including any of the following: a history of diarrhea, constipation, acid reflux, or abdominal pain as reported by the patient
* For women of childbearing age, effective contraception must be used before beginning CellCept or Myfortic, during therapy and 6 weeks after therapy has been discontinued (childbearing women should have a negative serum or urine pregnancy test within 1 week prior to starting CellCept or Myfortic therapy)

Exclusion Criteria:

* Recipients with any prior solid organ transplant (including kidney)
* Recipients receiving a concurrent solid organ (heart, liver, pancreas) or cell (islet, bone marrow, stem cell) transplant
* Recipient age is less than 18 years old or greater than 75 years old
* Recipients who are not African American (self-reported patients of Black African descent who live in the United States)
* Recipients on proton pump inhibitor therapy at the time of initial screening (pre-transplant to 2 days post-transplant)
* Recipients with a gastrointestinal bleed within the past three months
* Recipients who are pregnant or breast feeding
* Recipients with known human immunodeficiency virus (HIV) infection
* Allergy to any of the immunosuppressant medications
* Concurrent investigational medication
* Any medical or psychosocial condition, which, in the opinion of the investigators, would hinder compliance with the study requirements
* Inability or unwillingness of patient to provide informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2007-03; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roy Bloom, MD, Principal Investigator — University of Pennsylvania-Renal Electrolyte and Hypertension Division
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occured at the Hospital of the University of Pennsylvania March 2007-June 2010. Living donor kidney recipients were approached in clinic at pre-transplant visit (within 30 days or less of transplant. Recipients of deceased donor kidney transplants were approached inpatient at transplant or 2 days thereafter.
Pre-assignment Details: Patients were not randomized until they were transplanted.
Groups:
- Myfortic Comparator Group: Patients in this group will receive Myfortic (enteric-coated mycophenolate sodium) 180 mg tablets administered as 720mg (4 tablets) orally twice daily (adjusted for side effects as needed) in addition to immunosuppressants: Thymoglobulin (Rabbit antithymocyte globulin), Prograf (tacrolimus) or its generic equivalanet and corticosteroids.
- CellCept Comparator Group: Patients in this group will receive CellCept (mycophenolate mofetil) 250mg capsules administered as 1000mg (4 capsules) orally twice daily (adjusted for side effects as needed) in addition to immunosuppressants: Thymoglobulin (rabbit anti-thymocyte globulin) Prograf (tacrolimus) or its generic equivalent and corticosteroids.
Period: Overall Study
Arm/Group | Myfortic Comparator Group | CellCept Comparator Group
Started | 18 | 19
Consented to Pharmacokinetic Study | 11 | 10
Completed 0/2 PK Visits | 3 | 4
Completed 1/2 PK Visits | 1 | 1
Completed 2/2 PK Visits | 7 | 5
Completed | 16 | 15
Not Completed | 2 | 4
Not completed — Adverse Event | 2 | 2
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Myfortic Comparator Group: Patients in this group will receive Thymoglobulin (rabbit anti-thymocyte globulin) induction immunosuppression in combination with Myfortic (enteric-coated mycophenolate sodium), Prograf (tacrolimus) or its generic equivalent and corticosteroid immunosuppression
- CellCept Comparator Group: Patients in this group will receive Thymoglobulin (rabbit anti-thymocyte globulin) induction immunosuppression in combination with CellCept (mycophenolate mofetil) or its generic equivalent, Prograf (tacrolimus) or its generic equivalent and corticosteroid immunosuppression.
- Total: Total of all reporting groups
Arm/Group | Myfortic Comparator Group | CellCept Comparator Group | Total
Number analyzed (Participants) | 18 | 19 | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 19 | 37
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.9 (9.3) | 52.4 (13.0) | 50.3 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 13
  Male | 11 | 13 | 24
Region of Enrollment [Number; unit: participants]
  United States | 18 | 19 | 37

OUTCOME MEASURES:

1. Primary Outcome: Gastrointestinal Toxicity Due to Enteric Coated Mycophenolate Sodium or Mycophenolate Mofetil or Its Generic Equivalent Formulation Manufactured by Sandoz
Description: At 24 weeks, we assessed the number of patients at this timepoint who required permanent dose decrease or discontinuation of either enteric coated mycophenolate sodium or mycophenolate mofetil or its generic equivalent formulation manufactured by Sandoz related to gastrointestinal toxicity.
Time Frame: 6 months
Population: Based on the number of patients who were participating in the trial at that timepoint and had not withdrawn at 24 weeks
Measure: Number; unit: participants
Arm/Group | Myfortic Comparator Group | CellCept Comparator Group
Number analyzed (Participants) | 17 | 14
participants | 9 | 4
Statistical Analysis 1: Comparison: Myfortic Comparator Group vs CellCept Comparator Group; Sample size was arbitrarily determined as 40 patients (20 in the CellCept group and 20 in the Myfortic group) in this proof of concept study; Test type: Superiority; p = .29, Fisher Exact — A p value of less than 0.05 was considered statistically significant

2. Secondary Outcome: The Incidence of the Requirement of Full Dose Proton Pump Inhibitors in Patients on Enteric Coated Mycophenolate Sodium or Mycophenolate Mofetil or Its Generic Equivalent Manufactured by Sandoz
Description: If patients were not on any medications from a medication class known as H-2 antagonists, they were started on ranitidine 150 mg orally twice daily after transplant (with dose adjusted for renal function). Patients were excluded if they were on proton pump inhibitor at time of study screening, however some patients required addition of proton pump inhibitor post-study enrollment. If a patient had upper gastrointestinal side effects such as acid reflux unreleived on ranitidine therapy or nausea, they were switched to a proton pump inhibitor.
Time Frame: 6 months
Population: Based on number of patients participating in study at 6 months
Measure: Number; unit: participants
Arm/Group | Myfortic Comparator Group | CellCept Comparator Group
Number analyzed (Participants) | 17 | 14
participants | 3 | 1
Statistical Analysis 1: Comparison: Myfortic Comparator Group vs CellCept Comparator Group; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.39, Fisher Exact — A p value of less than 0.05 was considered statistically significant

3. Secondary Outcome: The Incidence of Intolerance (Defined as Transient Dose Reduction or Transient Discontinuation of Enteric Coated Mycophenolate Sodium or Mycophenolate Mofetil or Its Generic Equivalent Manufactured by Sandoz
Description: The incidence of intolerance was defined as transient dose reduction or transient discontinuation of enteric coated mycophenolate sodium or mycophenolate mofetil or its generic equivalent manufactured by Sandoz meaning doses could subsequently be resumed or increased back to original starting dose, once intolerance resolved.
Time Frame: 6 months
Population: Based on number of patients participating in the study at 6 months
Measure: Number; unit: participants
Arm/Group | Myfortic Comparator Group | CellCept Comparator Group
Number analyzed (Participants) | 17 | 14
participants | 1 | 0
Statistical Analysis 1: Comparison: Myfortic Comparator Group vs CellCept Comparator Group; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 1.0, Fisher Exact — A p value of less than 0.05 was considered statistically significant

4. Secondary Outcome: Gastrointestinal Symptom Rating Scale (GSRS) Score Changes From Baseline to 24 Weeks After Transplant in Patients on Enteric Coated Mycophenolate Sodium or Mycophenolate Mofetil or Its Generic Equivalent Manufactured by Sandoz
Description: The Gastrointestinal Symptom Rating Scale (GSRS) is a 15-item self-administered questionnaire to assess symptoms associated with common gastrointestinal (GI) disorders, and has been validated in renal transplant recipients. It uses a seven-graded Likert scale, where 1 represents the most positive option and 7 the most negative one and the patient grades symptoms based on the past 7 days. A score of ≥ 2 indicates the presence of GI symptoms. Higher values indicate more unfavorable conditions. The questionairre is divided into 5 sub-scales: diarrhea, indigestion, constipation, abdominal pain, and reflux and a mean score is calculated for each dimension. The lowest mean score possible for each dimension is 1 and the highest is 7. Patients completed a GSRS survey at baseline (pre-transplant to two days after transplant), and at weeks 1,4,12 and 24 after transplant.
Time Frame: baseline (pre-transplant to two days after transplant) and at 6 months after transplant.
Population: Patients who withdrew from the study before 24 weeks were excluded from this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Myfortic Comparator Group | CellCept Comparator Group
Number analyzed (Participants) | 17 | 14
Participants
  Worsening of GSRS Score pre-transplant-wk 24 | 4 | 4
  No Worsening of GSRS Score pre-transplant-wk 24 | 13 | 10
Statistical Analysis 1: Comparison: Myfortic Comparator Group vs CellCept Comparator Group; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 1.00, Fisher Exact — A p value of less than 0.05 was considered significant

5. Secondary Outcome: The Incidence of the Occurrence of Upper Gastrointestinal Symptoms Per GSRS Scale Ratings in Patients on Enteric Coated Mycophenolate Sodium or Mycophenolate Mofetil or Its Generic Equivalent Formulation Manufactured by Sandoz
Description: The Gastrointestinal Symptom Rating Scale (GSRS) is a 15-item self-administered questionnaire to assess symptoms associated with common gastrointestinal (GI) disorders, and has been validated in renal transplant recipients. It uses a seven-graded Likert scale, where 1 represents the most positive option and 7 the most negative one and the patient grades symptoms based on the past 7 days. A score of ≥ 2 indicates the presence of GI symptoms. Higher values indicate more unfavorable conditions. The questionairre is divided into 5 sub-scales: diarrhea, constipation, abdominal pain, indigestion and reflux and a mean score is calculated for each dimension. The lowest mean score possible for each dimension is 1 and the highest is 7. Patients completed a GSRS survey at baseline (pre-transplant to two days after transplant), and at weeks 1,4,12 and 24 post-transplant.
Time Frame: 6 months
Population: Any patient with mean GSRS subscale score >1 from dimensions: abdominal pain, indigestion, or reflux were considered to have upper GI symptoms.
Measure: Count of Participants; unit: Participants
Arm/Group | Myfortic Comparator Group | CellCept Comparator Group
Number analyzed (Participants) | 17 | 14
Participants
  Number of Participants with Upper GI symptoms | 8 | 11
  Number of Participants without Upper GI symptoms | 9 | 3
Statistical Analysis 1: Comparison: Myfortic Comparator Group vs CellCept Comparator Group; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.14, Fisher Exact — a p value of less than 0.05 was considered statistically significant

6. Secondary Outcome: The Incidence of the Occurrence of Lower Gastrointestinal Symptoms Per GSRS Scale Ratings in Patients on Enteric Coated Mycophenolate Sodium or Mycophenolate Mofetil or Its Generic Equivalent Manufactured by Sandoz
Description: The Gastrointestinal Symptom Rating Scale (GSRS) is a 15-item self-administered questionnaire to assess symptoms associated with common gastrointestinal (GI) disorders, and has been validated in renal transplant recipients. It uses a seven-graded Likert scale, where 1 represents the most positive option and 7 the most negative one and the patient grades symptoms based on the past 7 days. A score of ≥ 2 indicates the presence of GI symptoms. Higher values indicate more unfavorable conditions. The questionairre is divided into 5 sub-scales: diarrhea, constipation, abdominal pain, indigestion and reflux and a mean score is calculated for each dimension. The lowest mean score possible for each dimension is 1 and the highest is 7. Patients completed a GSRS survey at baseline (pre-transplant to two days after transplant), and at weeks 1,4,12 and 24 post-transplant. Patients who withdrew from the study only had data included up to the point of withdraw. No values were carried forward.
Time Frame: 6 months
Population: Any patient with a mean GSRS subscale score > 1 on dimensions constipation or diarrhea were considered to have lower GI symptoms.
Measure: Count of Participants; unit: Participants
Arm/Group | Myfortic Comparator Group | CellCept Comparator Group
Number analyzed (Participants) | 17 | 14
Participants
  Number of Participants with Lower GI symptoms | 8 | 9
  Number of Participants without Lower GI symptoms | 9 | 5
Statistical Analysis 1: Comparison: Myfortic Comparator Group vs CellCept Comparator Group; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.34, Chi-squared — A p value of less than 0.05 was considered statistically significant

7. Secondary Outcome: The Incidence of Rejection in Patients on Enteric Coated Mycophenolate Sodium or Mycophenolate Mofetil or Its Generic Equivalent Manufactured by Sandoz.
Description: All rejection episodes of the kidney transplant were proven by kidney transplant biopsy and were measured at 24 weeks for all patients still participating in the study at that timepoint.
Time Frame: 6 months
Population: Included any patient who experienced rejection while enrolled in the study up to 6 months post-transplant.
Measure: Number; unit: participants
Arm/Group | Myfortic Comparator Group | CellCept Comparator Group
Number analyzed (Participants) | 17 | 14
participants | 2 | 1
Statistical Analysis 1: Comparison: Myfortic Comparator Group vs CellCept Comparator Group; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = .51, Fisher Exact — A p-value of less than 0.05 was considered statistically significant

8. Secondary Outcome: Serum Creatinine in Patients on Enteric Coated Mycophenolate Sodium or Mycophenolate Mofetil or Its Generic Equivalent Manufactured by Sandoz
Description: Serum creatinine lab values were used as part of a measure of renal function at 24 weeks for any patient that was still participating in the study at this time-point.
Time Frame: 6 months
Population: Any patient with serum creatinine values available at 24 weeks
Measure: Mean (Standard Deviation); unit: serum creatinine mg/dL
Arm/Group | Myfortic Comparator Group | CellCept Comparator Group
Number analyzed (Participants) | 17 | 14
serum creatinine mg/dL | 1.9 (3.0) | 1.9 (0.9)
Statistical Analysis 1: Comparison: Myfortic Comparator Group vs CellCept Comparator Group; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.95, t-test, 2 sided — A p-value of less than 0.05 was considered statistically significant

9. Secondary Outcome: Modification of Diet and Renal Disease (MDRD) Measured Glomerular Filtration Rates in Patients on Enteric Coated Mycophenolate Sodium or Mycophenolate Mofetil or Its Generic Equivalent Manufactured by Sandoz
Description: Modification of Diet and Renal Disease (MDRD) Measured Glomerular Filtration Rates were used as part of a measure of renal function and measured at 24 weeks in patients who were still participating in the study at that point.
Time Frame: 6 months
Population: Any patient with Modification of Diet and Renal Disease (MDRD) Measured Glomerular Filtration Rates at 24 weeks was included in the analysis
Measure: Mean (Standard Deviation); unit: MDRD (mL/min/1.73m2)
Arm/Group | Myfortic Comparator Group | CellCept Comparator Group
Number analyzed (Participants) | 17 | 14
MDRD (mL/min/1.73m2) | 59.6 (22.5) | 54.8 (20.0)
Statistical Analysis 1: Comparison: Myfortic Comparator Group vs CellCept Comparator Group; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.57, t-test, 2 sided — The p value was not adjusted for multiple comparisons. A p-value of less than 0.05 was considered statistically significant

10. Secondary Outcome: Pharmacokinetics (Mycophenolic Acid Trough Levels) of Enteric Coated Mycophenolate Sodium or Mycophenolate Mofetil or Its Generic Equivalent Manufactured by Sandoz in a Sub-set of Patients
Description: Pharmacokinetics is the study of how a drug is absorbed and broken down in the body. Pharmacokinetics of enteric coated mycophenolate sodium and mycophenolate mofetil are measured by a level called mycophenolic acid level. Mycophenolic acid levels in this pharmacokinetic study were drawn starting in the morning at time zero (immediately prior to morning dose, also known as trough), then at 0.5, 1,1.5, 2, 2.5, 3,3.5,4,6, 8 and 12 hours post dose. Data was also dose-normalized (concentration was divided by dose).
Time Frame: 1 and 6 months
Population: Any participant who completed at least one pharmacokinetic studies was included in this analysis.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Myfortic Comparator Group | CellCept Comparator Group
Number analyzed (Participants) | 8 | 6
mg/L
  Mycophenolic Acid Trough (mg/L) at week 4 | 2.4 (1.6) | 1.9 (1.3)
  Mycophenolic Acid Trough(mg/L) at week 24: number analyzed (Participants) | 7 | 5
  Mycophenolic Acid Trough(mg/L) at week 24 | 1.9 (1.5) | 1.5 (1.1)
Statistical Analysis 1: Comparison: Myfortic Comparator Group vs CellCept Comparator Group; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.45, Kruskal-Wallis — This represents p value for week 4 data. A p value of less than 0.05 was considered significant
Statistical Analysis 2: Comparison: Myfortic Comparator Group vs CellCept Comparator Group; Sample size was arbitrarily determined as 40 patients (20 in CellCept group and 20 in the Myfortic group) in this proof of concept study; Test type: Superiority; p = 0.58, Kruskal-Wallis — This represents p value for week 24 data. A p value of less than 0.05 was considered significant

11. Secondary Outcome: Pharmacokinetics (Mycophenolic Acid Maximum Concentration) of Enteric Coated Mycophenolate Sodium or Mycophenolate Mofetil or Its Generic Equivalent Manufactured by Sandoz in a Sub-set of Patients
Description: Pharmacokinetics is the study of how a drug is absorbed and broken down in the body. Pharmacokinetics of Enteric-Coated Mycophenolate Sodium or Mycophenolate Mofetil are measured by a level called mycophenolic acid level. Mycophenolic acid levels in this pharmacokinetic study were drawn starting in the morning at time zero (immediately prior to morning dose, also known as trough), then at 0.5, 1,1.5, 2, 2.5, 3,3.5,4,6, 8 and 12 hours post dose. Data was also dose-normalized (concentration was divided by dose).A mycophenolic acid drawn at the peak level is called C Max or maximum concentration.
Time Frame: 1 and 6 months
Population: Any participant who completed at least one pharmacokinetic studies was included in this pharmacokinetic analyses.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Myfortic Comparator Group | CellCept Comparator Group
Number analyzed (Participants) | 8 | 6
mg/L
  Mycophenolic Acid C max (mg/L) at week 4 | 4.3 (1.5) | 10.5 (4.1)
  Mycophenolic Acid C max (mg/L) at week 24: number analyzed (Participants) | 7 | 5
  Mycophenolic Acid C max (mg/L) at week 24 | 6.4 (3.5) | 13.9 (6.0)
Statistical Analysis 1: Comparison: Myfortic Comparator Group vs CellCept Comparator Group; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.012, Kruskal-Wallis — This p value is for data at week 4. A p value of less than 0.05 was considered significant
Statistical Analysis 2: Comparison: Myfortic Comparator Group vs CellCept Comparator Group; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.046, Kruskal-Wallis — This p value was for data at week 24. A p value of less than 0.05 was considered significant

12. Secondary Outcome: Pharmacokinetics (Mycophenolic Acid Area Under the Curve) of Enteric Coated Mycophenolate Sodium or Mycophenolate Mofetil or Its Generic Equivalent Manufactured by Sandoz in a Sub-set of Patients
Description: Pharmacokinetics is the study of how a drug is absorbed and broken down in the body. Pharmacokinetics of Enteric-Coated Mycophenolate Sodium or Mycophenolate Mofetil are measured by a level called mycophenolic acid level. Mycophenolic acid levels in this pharmacokinetic study were drawn starting in the morning at time zero (immediately prior to morning dose, also known as trough), then at 0.5, 1,1.5, 2, 2.5, 3,3.5,4,6, 8 and 12 hours post dose. Data was also dose-normalized (concentration was divided by dose). A mycophenolic acid area under the curve value, also known as AUC represents drug exposure.
Time Frame: 1 and 6 months
Population: Any participant who completed at least one pharmacokinetic studies was included in this pharmacokinetic analyses.
Measure: Mean (Standard Deviation); unit: mg*hr/L
Arm/Group | Myfortic Comparator Group | CellCept Comparator Group
Number analyzed (Participants) | 8 | 6
mg*hr/L
  Mycophenolic Acid AUC (mg*hr/L) at week 4 | 23.9 (10.9) | 33.8 (18.4)
  Mycophenolic Acid AUC (mg*hr/L) at week 24 | 21.1 (11.7) | 42.4 (33.2)
Statistical Analysis 1: Comparison: Myfortic Comparator Group vs CellCept Comparator Group; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.27, Kruskal-Wallis — p value represents data for week 4. A p value of less than 0.05 was considered significant
Statistical Analysis 2: Comparison: Myfortic Comparator Group vs CellCept Comparator Group; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.23, Kruskal-Wallis — p value represents data for week 24. A p value of less than 0.05 was considered significant

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Myfortic Comparator Group | CellCept Comparator Group
Serious Adverse Events (participants affected / at risk) | 18/18 | 19/19
Other Adverse Events (participants affected / at risk) | 18/18 | 17/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Myfortic Comparator Group (N=18) | CellCept Comparator Group (N=19)
graft dysfunction due to rejection (Renal and urinary disorders) | 1 (2) | 1 (1)
non-infectious related diarrhea (Gastrointestinal disorders) | 2 (2) | 3 (3)
lymphocele (Injury, poisoning and procedural complications) | 0 (0) | 2 (4)
graft failure due to antibody mediated rejection (Renal and urinary disorders) | 1 (1) | 0 (0) — Occurred during 30 day safety follow-up period when patient was found to be non-adherent with immunosuppression. Antibody mediated rejection was considered non-reversible and patient progressed to graft failure.
dialysis fistula thrombosis (Vascular disorders) | 1 (1) | 0 (0) — Patient had dialysis fistula thrombosis during treatment for antibody mediated rejection that progressed to graft failure in 30 day safety follow-up period due to non-adherence.
urinary leak post renal transplant (Renal and urinary disorders) | 0 (0) | 1 (1)
diabetic complications (Metabolism and nutrition disorders) | 1 (1) | 4 (4)
dehydration (Renal and urinary disorders) | 0 (0) | 1 (1)
graft dysfunction not found to be related to rejection (Renal and urinary disorders) | 3 (4) | 6 (9) — causes included acute tubular necrosis, chronic allograft nephropathy, recurrent focal segmental glomerulosclerosis
anemia managed during hospitalization (Renal and urinary disorders) | 2 (2) | 3 (3)
failure to thrive (Renal and urinary disorders) | 0 (0) | 1 (1)
high potassium (hyperkalemia) requiring hospitalization for management (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
cervical arthritis and related neuropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) — patient redmitted for dehydration and vomiting
thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Bacterial infections (Infections and infestations) | 6 (7) | 5 (5) — infection
Viral infections (Infections and infestations) | 1 (1) | 2 (2) — infection
wound seroma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — wound seroma
heart complications (Cardiac disorders) | 2 (2) | 1 (1) — non-sustained ventricular tachycardia, pericardial effusion, myocardial infarction
wound complications (Surgical and medical procedures) | 1 (1) | 0 (0) — wound vac placement
recurrence of renal disease (Renal and urinary disorders) | 0 (0) | 1 (1) — recurrent primary disease FSGS
drug induced rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — thought to be related to rabbit anti-thymocyte globulin induction
Leg pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — unrelated to vascular complications or infection
high blood pressure (Cardiac disorders) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Myfortic Comparator Group (N=18) | CellCept Comparator Group (N=19)
Muscle cramps (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Heartburn (Gastrointestinal disorders) | 3 (3) | 5 (5)
Diabetic Complications (Endocrine disorders) | 4 (4) | 0 (0) — worsening pre-transpalnt diabets blood sugar control
superior vena cava syndrome (Vascular disorders) | 1 (1) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 7 (7) | 6 (6)
bacterial infection not requiring hospitalization (Infections and infestations) | 3 (4) | 0 (0) — urinary tract infection
soft stools without diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1)
high potassium (hyperkalemia) not requiring hospitalization (Metabolism and nutrition disorders) | 5 (5) | 5 (5)
urinary retention not requiring hospitalization (Renal and urinary disorders) | 1 (1) | 1 (1)
low white blood cell count (leukopenia) (Blood and lymphatic system disorders) | 4 (4) | 3 (3)
accidental anti-anxiety pill overdose not requiring inpatient hospitalization (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
increased bowel movement frequency (Gastrointestinal disorders) | 1 (1) | 0 (0)
delayed graft function of renal transplant (Renal and urinary disorders) | 9 (9) | 8 (8)
nausea (Gastrointestinal disorders) | 1 (1) | 2 (2) — nausea resulted in subsequent weight loss not requiring hospitalization in one cellcept patient and associated also with vomiting in one patient on cellcept
low platelet count (thrombocytopenia) (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
nephrotic range protein in urine (proteinuria) (Renal and urinary disorders) | 0 (0) | 1 (1)
blurry vision (Eye disorders) | 0 (0) | 1 (1) — did not require any intervention and resolved on own
low red blood cell count (anemia) (Blood and lymphatic system disorders) | 5 (5) | 3 (3)
shortness of breath and fluid related weight gain not requiring hospitalization (Cardiac disorders) | 2 (2) | 0 (0)
hemmorhoids (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
back pain after fall on ice (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
viral cold infection (Infections and infestations) | 2 (2) | 0 (0) — resolved on its own without treatment
hip-pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) — no source found in one patient and other patient had history of pre-transplant avascular necrosis
tertiary hyperparathyroidism (Endocrine disorders) | 1 (1) | 0 (0) — treated with oral medication as outpatient
root canal (Surgical and medical procedures) | 1 (1) | 0 (0)
high hemoglobin (Blood and lymphatic system disorders) | 1 (1) | 1 (1) — treated with outpatient phlebotomy
mild increase in liver function tests (transaminitis) (Hepatobiliary disorders) | 1 (1) | 0 (0) — patient had history of pre-transplant hepatitis B infection
hypoglycemia (low blood sugars) (Endocrine disorders) | 1 (1) | 0 (0) — patient was using sliding scale for elevated blood sugars but experienced hypoglycemia-resolved upon stopping insulin and patient did not need any further therapy
bled through non-functioning dialysis graft not requiring inpatient hospitalization (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
bk virus infection (Infections and infestations) | 1 (1) | 2 (2) — was BKV nephropathy in one myfortic patient
high cholesterol (hyperlipidemia) (Cardiac disorders) | 0 (0) | 1 (1) — Patient was on maximum statin dose. Symptoms resolved with diet, exercise and decreased prednisone dose.
abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) — symptoms improved over time without any specific treatment
skin itching thought to be related to dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
metabolic acidosis (Renal and urinary disorders) | 1 (1) | 0 (0) — treated as outpatient with oral bicarbonate and resolved
blood in urine and mild transplant rejection (Renal and urinary disorders) | 1 (1) | 0 (0) — treated as outpatient with pulse steroid doses
renal dysfunction and edema (Renal and urinary disorders) | 1 (1) | 1 (1) — found to be related to SVC in 30+ day follow-up in MMF group patient
low phosphorous (Metabolism and nutrition disorders) | 1 (1) | 0 (0) — corrected with diet
bowel urgency (Gastrointestinal disorders) | 1 (1) | 0 (0)
unilateral lower leg swelling (General disorders) | 1 (1) | 0 (0) — not transplant related and negative for deep vein thrombosis
low potassium (Metabolism and nutrition disorders) | 1 (1) | 0 (0) — resolved with change in diet
neck itching (Immune system disorders) | 1 (1) | 0 (0) — patient thought symptoms may be related to allergy and resolved with otc medication product change.
muscle leg pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — resolved with prescription muscle relaxant
ongoing high blood pressure (Cardiac disorders) | 1 (1) | 1 (1) — ongoing high blood pressure on medications
hot flashes (General disorders) | 1 (1) | 0 (0)
lymphocele or seroma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — stable on outpatient ultrasound

LIMITATIONS AND CAVEATS:
Limitations of our study include small sample size and patient drop out-though not significantly different between the MMF and EC-MPS groups and limited follow-up

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No